CLINICAL TRIAL: NCT03153826
Title: Determinants of Lower Limb Muscle Atrophy Induced During an Hospitalization for Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Determinants of Lower Limb Muscle Atrophy Induced During an Hospitalization for Exacerbation of COPD
Acronym: AMI-EX-BPCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient recruitment
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9774
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Exacerbation Copd; Muscle Atrophy
Keywords: COPD Exacerbation; Muscle atrophy; Inflammation; Oxidative stress
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other)
  Interventions: Other: Comparison of clinical and biological characteristics of patients

INTERVENTIONS:
Other: Comparison of clinical and biological characteristics of patients — Comparison of clinical and biological characteristics of patients with less variation in muscle mass (evaluated by CSARF) compared to patients with greater variation during an hospitalization for COPD exacerbation

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by persistent airway obstruction and inflammatory response of the lungs and bronchi. Episodes of exacerbations contribute to increase the severity and prognosis of the disease. Muscle dysfunction (loss of strength and muscle mass) is one of comorbidities affecting 30% to 60% of patients and playing a key role in their prognosis. Indeed, several studies have shown muscle weakness during hospitalization for exacerbation of COPD by measure of maximal voluntary contraction of quadriceps (MVCQ), but the results are variable from one patient to another. Moreover, no study was interested in the change of muscle mass in patients hospitalized for an exacerbation of COPD. Several mechanisms have been mentioned but not demonstrated: systemics factors (initial amyotrophy, inflammation, oxidative stress, corticotherapy, hypoxia…) but also physical inactivity. In this context, identifying factors associated with the onset of muscle weakness during hospitalization for exacerbation of COPD is a necessary step to better understand the mechanisms and consider a personalized therapeutic approach that can improve the functional and clinical prognosis of disease.

The primary outcome is to identify the clinical and biological determinants associated with the onset of amyotrophy (Measure by ultrasound of sectional area of the Rectus Femoris, CSARF), during hospitalization for exacerbation of COPD. The secondary outcome is to identify the clinical and biological determinants associated with the onset of MVCQ decrease, during hospitalization for exacerbation of COPD.

120 patients hospitalized for exacerbation of COPD will be recruited in two hospitals (CHU Montpellier - CHU Grenoble, FRANCE). The measures of CSARF and MVCQ are carried out on the second, fifth, eighth day of hospitalization, on discharge and on the sixtieth day after hospitalization. A blood test will be performed on the second day of hospitalization to explore different markers of inflammation and oxydative stress. Moreover, to quantify the level of physical activity (number of steps), each patient will carry a pedometer throughout the duration of hospitalization.

At the end of protocol, two groups will be made from the median of CSARF : patients with a small reduction in CSARF compared to patients with a greater reduction in SSRF between the second and eighth days of hospitalization (or between the second day of hospitalization and discharge). Then clinical (comorbidities, severity disease, initial weakness, initial amyotrophy, usual physical activity before hospitalization, treatment, exacerbation number in the previous year…) and biological (markers of inflammation and oxydative stress) determinants were compared between the two groups.

Thus, the identification of the determinants associated with the onset of amyotrophy induced during exacerbation of COPD will guide research for exploration of physiopathological mechanisms of this muscular dysfunction in the exacerbation of COPD as well as to identify a personalized support.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 40 to 85 years
* COPD patients : FEV1/FVC < 70% pred
* Hospitalization for COPD exacerbation : increased respiratory symptoms over two consecutive days with at least one major symptom (dyspnea, increased sputum volume or purity) associated with another major symptom or minor symptom (sibilant, cold, sore throat or cough)

Exclusion criteria:

* Concomitant cardiac event
* Tracheal intubation
* Chronic respiratory disease other than COPD
* Disease of locomotor apparatus, neurological or psychiatrics comorbidities

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical and biological characteristics of patients | Second day after hospitalization and discharge
  Comparison of clinical and biological characteristics of patients with less variation in muscle mass (evaluated by CSARF) compared to patients with greater variation during an hospitalization for COPD exacerbation
Comparison of clinical and biological characteristics of patients | Fifth day after hospitalization and discharge
  Comparison of clinical and biological characteristics of patients with less variation in muscle mass (evaluated by CSARF) compared to patients with greater variation during an hospitalization for COPD exacerbation
Comparison of clinical and biological characteristics of patients | Eigth day after hospitalization and discharge
  Comparison of clinical and biological characteristics of patients with less variation in muscle mass (evaluated by CSARF) compared to patients with greater variation during an hospitalization for COPD exacerbation

SECONDARY OUTCOMES:
Comparison of clinical and biological characteristics | Second, fifth, and eighth day after hospitalization and discharge
  Comparison of clinical and biological characteristics of patients with less variation in maximal voluntary contraction of quadriceps (MVCQ) compared to patients with greater variation during an hospitalization for COPD exacerbation

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital Arnaud de Villeneuve Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No